CLINICAL TRIAL: NCT04132284
Title: Pilot Randomized Controlled Trial of a DBT-based Parenting Intervention
Brief Title: DBT-Based Parenting Intervention for Parents of Youth at Risk for Suicide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michele Berk, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 50613
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Adolescent - Emotional Problem; Suicide and Self-harm; Parenting
MeSH Terms: conditions — Suicide; Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT IOP plus DBT PI (Experimental): Standard Dialectical Behavior Therapy (DBT) delivered in the context of an intensive outpatient program (DBT IOP) for adolescents plus an 8-10 session DBT-based parenting intervention (DBT PI)
  Interventions: Behavioral: DBT-Based Parenting Intervention
- DBT IOP alone (Active Comparator): No parenting intervention provided beyond what is part of the DBT IOP treatment as usual.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: DBT-Based Parenting Intervention — The intervention will consist of 8-10 individual parent sessions, to be completed within one week after the teen completes the IOP program. Sessions will be 1 hour in length and will be offered weekly. Therapists may see parents more than once a week if needed, as long as the total number of sessions does not exceed 10. Sessions will follow the standard agenda used for DBT skills training: 1) mindfulness practice, 2) homework review, 3) teaching of a new skill; 4) practice of the new skill; and 5) assignment of new homework (Linehan, 1993). The intervention will utilize the Middle Path module of the DBT Skills Manual for Adolescents (Rathus & Miller, 2015), which was created by the developers of DBT for adolescents and includes both instructions for therapists and handouts for clients.
  Arms: DBT IOP plus DBT PI
Behavioral: Treatment as Usual — No parenting intervention provided beyond standard practices in DBT IOP program.
  Arms: DBT IOP alone

SUMMARY:
The purpose of the present study is to conduct a pilot randomized clinical trial (RCT) of an 8-10 session DBT-based parenting intervention (DBT PI) plus standard Dialectical Behavior Therapy delivered in the context of an intensive outpatient program (DBT IOP) to DBT IOP alone. The long term goal of the research is to determine if augmenting standard DBT with additional parenting intervention improves youth treatment response on suicide-related outcomes (i.e., suicidal ideation, non-suicidal self-injury and suicide attempts). The goal of this pilot RCT is to collect preliminary data needed for a larger RCT, including feasibility, acceptability, safety, tolerability, engagement of the presumed mechanism of change (changes in parent emotions and behaviors) and signal detection of any changes in youth suicide-related outcomes.

DETAILED DESCRIPTION:
The present study is a pilot RCT of a DBT parenting intervention (DBT PI). The investigators will enroll N = 40 pairs of youth and parents enrolled in a DBT intensive outpatient program that delivers standard DBT (DBT IOP). This program, called the RISE program, is jointly run by Stanford and Children's Health Council (CHC). CHC is a community mental health clinic located in Palo Alto and is where the IOP is housed. All research procedures will be conducted by Stanford faculty and staff. Parents and youth who provide informed consent will be randomly assigned to receive the DBT PI + DBT IOP or DBT IOP only. Parents assigned to the DBT PI + DBT IOP will be offered 10 sessions of DBT-based parenting interventions. Youth will participate in study assessments only and will not receive additional treatment as part of the study (i.e., they will receive DBT IOP only). Study participation is optional and will not impact the family's ability to participate in the DBT IOP. Youth will be enrolled in the IOP program as part of standard clinical practices, regardless of whether or not they choose to participate in the study. Assessments will be conducted at baseline, 3-month follow-up (end of DBT IOP program) and 6 month follow-up. Both parents will be encouraged to take part in the intervention, however; the participation of only one parent will be required. The intervention will consist of 8-10 individual parent sessions, to be completed within one week after the teen completes the IOP program. Sessions will be 1 hour in length and will be offered weekly. Therapists may see parents more than once a week if needed, as long as the total number of sessions does not exceed 10. Sessions will follow the standard agenda used for DBT skills training: 1) mindfulness practice, 2) homework review, 3) teaching of a new skill; 4) practice of the new skill; and 5) assignment of new homework (Linehan, 1993). The intervention will utilize the Middle Path module from the DBT Skills Manual for Adolescents (Rathus & Miller, 2015), which was created by the developers of DBT for adolescents and includes both instructions for therapists and handouts for clients.

ELIGIBILITY:
Inclusion Criteria:

1) youth is enrolled in CHC-Stanford RISE program; 2) youth and parent are willing to participate, and 3) youth and parent speak English.

Exclusion Criteria:

1) the youth or parent has a psychiatric or medical condition that would interfere with their ability to participate in study assessments and/or treatment (such as acute psychosis, neurological impairment, malnutrition due to severe anorexia).

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Number of Youth Self-Harm Episodes | 6 months
Youth Suicidal Ideation | 6 months

SECONDARY OUTCOMES:
Parent Emotion Dysregulation | 6 months
Parent Depressive Symptoms | 6 months
Parent Caregiver Strain | 6 months
Family Conflict | 6 months
Family Functioning McMaster Family Assessment Device | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No